CLINICAL TRIAL: NCT03662490
Title: Correlation Between Clinical Signs and High-resolution Manometry Data in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-54
Record Dates: First submitted 2018-09-06; First posted 2018-09-07 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Oesophageal Motility Disorder
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Patient who performed a High resolution oesophageal manometry (HRM) for the diagnosis of oesophageal motility disorder.
  Interventions: Device: High resolution oesophageal manometry

INTERVENTIONS:
Device: High resolution oesophageal manometry — High resolution oesophageal manometry (HRM) is the gold standard for the diagnosis of oesophageal motility disorder.

SUMMARY:
High resolution oesophageal manometry (HRM) is the gold standard for the diagnosis of oesophageal motility disorder.

Standard esophageal manometry has been replaced since 2000 by high resolution manometry. This one allows a more precise study with a spatio-temporal representation of the esophageal pressure values as well as an easier realization with in particular a better tolerance of the examination which is important in pediatrics.

Over a period of 10 years only a dozen studies were conducted in children. No study to date has evaluated the global place of MHR in current practice in children across all indications.

The indications that lead to the realization of a manometry in children are given by some experts but there is currently no clinical study to define the sensitivities, specificity and predictive values of clinical symptoms leading to the completion of this examination and endoscopic signs found upstream.

In addition, the link between certain underlying conditions and the manometric result has never been evaluated.

II / Objective: The objective of our study is to calculate the sensitivity, the specificity and the predictive values of each clinical and endoscopic sign according to the manometric result found and this by age group. The goal is to better define the predictive signs of the selected manometric diagnoses and therefore the indications to remember in the child.

III / Methodology:

Bi-centric retrospective collection of data on patient records in Marseille and Lille. Collection dates: from 2012 (beginning of high resolution manometry in Marseille and Lille) to December 2016.

The clinical and endoscopic signs selected will be decided a priori by an expert committee consisting of 2 adult gastroenterologists specializing in manometry, 1 pediatrician specialist in manometry, and 3 gastro-pediatricians.

Inclusion Criteria: All minor patients (<18 years old) referred for 1 st high-resolution manometry (or 2 nd or more examination if performed in the presence of a new symptom).

Number of subjects planned: all the patients who had a manometry (about 300 patients) over the given period

DETAILED DESCRIPTION:
High resolution oesophageal manometry (HRM) is the gold standard for the diagnosis of oesophageal motility disorder.

Standard esophageal manometry has been replaced since 2000 by high resolution manometry. This one allows a more precise study with a spatio-temporal representation of the esophageal pressure values as well as an easier realization with in particular a better tolerance of the examination which is important in pediatrics.

Over a period of 10 years only a dozen studies were conducted in children. They focused on the technical aspects of the realization but especially of the interpretation of the examination or on specific pathologies well described: the atresia of the esophagus and achalasia. As a result, no study to date has evaluated the global place of MHR in current practice in children across all indications.

The indications that lead to the realization of a manometry in children are given by some experts but there is currently no clinical study to define the sensitivities, specificity and predictive values of clinical symptoms leading to the completion of this examination and endoscopic signs found upstream.

In addition, the link between certain underlying conditions and the manometric result has never been evaluated.

II / Objective: The objective of our study is to calculate the sensitivity, the specificity and the predictive values of each clinical and endoscopic sign according to the manometric result found and this by age group. The goal is to better define the predictive signs of the selected manometric diagnoses and therefore the indications to remember in the child.

III / Methodology:

Bi-centric retrospective collection of data on patient records in Marseille and Lille. Collection dates: from 2012 (beginning of high resolution manometry in Marseille and Lille) to December 2016.

The clinical and endoscopic signs selected will be decided a priori by an expert committee consisting of 2 adult gastroenterologists specializing in manometry, 1 pediatrician specialist in manometry, and 3 gastro-pediatricians.

Inclusion Criteria: All minor patients (<18 years old) referred for 1 st high-resolution manometry (or 2 nd or more examination if performed in the presence of a new symptom).

Number of subjects planned: all the patients who had a manometry (about 300 patients) over the given period

ELIGIBILITY:
Inclusion Criteria:

* All minor patients (<18 years old)
* Referred for 1 st high-resolution manometry (or 2 nd or more examination if performed in front of a new symptom).

Exclusion Criteria:

* Patients for whom the examination was a control of a previous examination.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All minor patients (<18 years old) referred for 1 st high-resolution manometry (or 2 nd or more examination if performed in front of a new symptom).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
number of clinical sign | one week
  Symptoms include: Dysphagia, Swallowing Disorders, Food Blockages, Oral Disorders, Vomiting, GERD, Anorexia, Weight Loss, Belching, Respiratory Exacerbations, and Back Sternal Pain.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France